CLINICAL TRIAL: NCT05955482
Title: PROMISE: Pragmatic Assessment of the NuvoAir Clinical Service in the Management of Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Pragmatic Assessment of the NuvoAir Clinical Service in the Management of Patients With Chronic Obstructive Pulmonary Disease
Acronym: PROMISE
Status: Active, not recruiting | Type: Observational
Sponsor: NuvoAir Medical PC (Industry)
Responsible Party: Sponsor
Other Study IDs: 50M16FSHP
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: COPD; Comorbidities and Coexisting Conditions
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NuvoAir Clinical service: Patients with COPD receiving usual care plus NuvoAir clinical services.
  Interventions: Other: NuvoAir Clinical Service
- Standard Care: Propensity matched controls with COPD who receive usual care.

INTERVENTIONS:
Other: NuvoAir Clinical Service — The NuvoAir clinical service offers comprehensive monitoring of health parameters and patient-reported outcomes as well as personalized clinical and behavioral interventions tailored to the patients' unique needs and their clinical risk. Furthermore, it involves virtual interaction with a NuvoAir Coach who provides guidance and assistance in navigating and utilizing the service. A dedicated NuvoAir care coordinator is available to offer self-management support and educational resources, aiming to enhance the management of COPD and other comorbidities. In situations where patients encounter new or worsening symptoms, the NuvoAir clinical team is accessible to provide medical intervention, advice and triage as required.
  Groups: NuvoAir Clinical service

SUMMARY:
This is a 12 month study of up to 500 people with COPD to determine if the NuvoAir clinical service leads to lower rates of severe COPD exacerbations, hospitalizations, emergency room visits, and total cost of care compared to a similar group that doesn't receive care from the NuvoAir clinical service.

DETAILED DESCRIPTION:
Description: The program will be a virtual (decentralized), pragmatic evaluation of an implementation of the NuvoAir Clinical service for patients with COPD residing in the United States of America and who are enrolled with one or more health insurers or providers supporting the program. The evaluation will be organized around two cohorts; Patients with an ICD10 code for COPD (in the health insurer's or provider's database);

* Who use the NuvoAir Clinical service vs those
* Who undergo standard care (matched control - no intervention)

Each patient in the NuvoAir cohort will receive their routine clinical care from their primary care provider with the addition of the NuvoAir Clinical service. The NuvoAir Clinical service offers comprehensive monitoring of health parameters and patient-reported outcomes as well as personalized clinical and behavioral interventions tailored to the patients' unique needs and their clinical risk. Furthermore, it involves virtual interaction with a NuvoAir Coach who provides guidance and assistance in navigating and utilizing the service. A dedicated NuvoAir care coordinator is available to offer self-management support and educational resources, aiming to enhance the management of COPD and other comorbidities. In situations where patients encounter new or worsening symptoms, the NuvoAir clinical team is accessible to provide medical intervention, advice and triage as required.

Each patient in the standard care cohorts will receive their routine clinical care from their healthcare provider as usual. Only anonymized data that is usually collected by their health insurer or provider will be subject to analysis, no additional data will be collected for the standard care cohort.

NuvoAir and standard care cohorts will be matched on the basis of age, gender, disease severity (ICD10 code for COPD with a severe exacerbation of COPD in the previous 12 months), geographic place and period of entry into the program. The program period will include 1 year of active participation (for NuvoAir users) followed by 1 year of follow-up using health insurer or provider records.

Objectives: To determine if use of the NuvoAir clinical service results in a lower rate and number of moderate and severe exacerbations of COPD, lower readmissions due to COPD exacerbation within a 30-day period following a COPD exacerbation, lower days in hospital and lower healthcare costs compared with the matched cohorts of standard care patients who do not use the NuvoAir clinical service. To determine if use of the NuvoAir results in reduced readmissions due to COPD during the 30-day period following an exacerbation, improved health status and improved adherence compared with prior to the program/baseline.

ELIGIBILITY:
Inclusion Criteria:

Have COPD, including emphysema and chronic bronchitis, per relevant COPD diagnostic codes in the past 2 years

* Are age ≥30 years
* Have access to a smartphone, cell phone, or landline telephone

Exclusion Criteria:

Do not have serious medical illness that would interfere with cooperation or understanding of instructions, including terminal illness, active substance abuse, or unstable mental illness or psychiatric condition

* Does not have severe uncompensated heart failure, acute cor pulmonale, clinically unstable pulmonary embolism, history of syncope related to forced expiration/cough, cerebral aneurysm, presence of pneumothorax.
* Is not pregnant or known intention to become pregnant within 12 months

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A propensity matched comparison group will be selected from the same insured population (Security Health Plan of Wisconsin): Patients with COPD of comparable COPD severity, age, gender from the same region and type of health insurance (Medicare Advantage).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Moderate & Severe Exacerbations | 12 months
  Rate of moderate and severe exacerbations of COPD, measured by the health insurer or provider's records.

SECONDARY OUTCOMES:
Readmissions | 30 days post admission
  Rate of hospital readmission in 30 days following COPD related hospitalization
Hospital days | 12 months
  Median number of hospital days
Cost of care | 12 months
  Total cost of care as measured by insurer claims data

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey VanWormer, PHD, Principal Investigator — Marshfield Clinic
Locations (1):
- Marshfield Clinic Research Institute, Marshfield, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No